CLINICAL TRIAL: NCT05826080
Title: The Cross-sectional Study and Longitudinal Study of the the Value of Adrenocorticotrophic Hormonestimulation in Adrenal Vein Sampling
Brief Title: Effect of Adrenocorticotropic Hormone Stimulation During Adrenal Vein Sampling in Primary Aldosteronism
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other)
Responsible Party: Sponsor
Other Study IDs: lp2023
Record Dates: First submitted 2023-04-11; First posted 2023-04-24 (Actual); Last update posted 2023-04-24 (Actual); Status verified 2022-10

CONDITIONS: Primary Aldosteronism; Aldosterone-Producing Adenoma; Idiopathic Hyperaldosteronism
Keywords: Primary aldosteronism; Adrenal vein sampling; Adrenocorticotrophic hormone; Selectivity index; Lateralization index; prognosis
MeSH Terms: conditions — Hyperaldosteronism; Adrenocortical Adenoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- operative group: Procedure/Surgery:Adrenal Vein Sampling;Adrenalectomy

SUMMARY:
The purpose of our research is to evaluate the value of ACTH stimulation in AVS especially in lateralization is still controversial.

DETAILED DESCRIPTION:
Primary aldosteronism (PA) is thought to be the most common secondary endocrine form of hypertension. A recent published study revealed that the prevalence of PA in patients with newly diagnosed hypertension in China was at least 4%. Compared with patients with essential hypertension with similar blood pressure, patients with PA have significantly higher atrial fibrillation, myocardial infarction, heart failure, stroke, deterioration of renal function and all-cause mortality. Therefore, early and systematic implementation of effective surgical or medical treatment is essential to prevent or reverse the excess vascular events and mortality of these patients.

Adrenal venous sampling (AVS) is key for reliable subtype identification recommended by different guidelines and consensus statements. However, AVS is a complex, technically challenging and expensive procedure, requiring proficient and dedicated interventional radiologists. More importantly, the standardised procedure and method of AVS have not been unified10. Adrenocorticotropic hormone (ACTH) infusion is employed by many centers to maximize the gradient in cortisol from the adrenal vein to the inferior vena cava, and to maximize aldosterone secretion from an aldosterone-producing adenomas (APA) and thus avoid the risk of sampling during a relatively quiescent phase of aldosterone secretion. There is no debate that ACTH stimulation increases the selectivity index (SI) and, therefore, greatly increases the likelihood of successful AVS. However, the effect of ACTH stimulation on the lateralization index (LI) is controversial, with several studies reporting a reduction in the proportion of lateralized AVS results and, therefore, of surgically treatable patients. Hitherto, most of the studies on the value of using ACTH stimulation in AVS are retrospective studies with a small sample size, or multi-center studies with ununified methods of ACTH stimulation and evaluation standards of results. Therefore, there are obvious heterogeneity in the results and the value of evidence is limited.

In this prospective study, we analyzed the SI and LI in simultaneous bilateral AVS at baseline and after ACTH stimulation in our center, and further estimated the prognosis of patients underwent adrenalectomy with different cut-off points of LI after ACTH stimulation. Present study will provide novel evidence for the value of ACTH stimulation in AVS and improve AVS procedure.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed as primary aldosteronism.
2. AVS was performed and conservative treatment or adrenalectomy was performed according to the results.
3. Regular follow-up was performed.

Exclusion Criteria:

1. Adrenal function evaluation suggests that it is complicated with hypercortisolism, subclinical hypercortisolism and pheochromocytoma.
2. Familial aldosteronism.
3. .Adrenal mass is considered to be malignant, or pathology suggests adrenocortical carcinoma.
4. .Complicated with severe infection, respiratory and circulatory failure, advanced tumor, severe. hepatic and renal insufficiency, neurological, psychiatric and immune deficiency diseases.
5. .Drugs: discontinuation of β-receptor inhibitors, angiotensin converting enzyme inhibitors, angiotensin Ⅱ receptor blockers, thiazide diuretics < 2 weeks, aldosterone receptor antagonists < 4 weeks.
6. .Pregnant and lactating women.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: primary aldosteronism patients
Sampling Method: Probability Sample
Enrollment: 59 (Estimated)
Dates: Start 2021-09-01 (Actual); Primary Completion 2023-10-01 (Estimated); Study Completion 2024-09-01 (Estimated)

PRIMARY OUTCOMES:
Participants' personal information | 1 day
  Self-reported information (the cause of discovering adrenal adenoma）
Physical assessments | 1 day
  BMI(body mess index) in kg/m^2
Screening test of primary aldosteronism（Supine standing test） | 1 day
  plasma aldosterone concentration in the supine position and standing position
Screening test of primary aldosteronism（Supine standing test） | 1 day
  plasma renin concentration in the supine position and standing position
Confirmatory test of primary aldosteronism（Captopril test） | 1 day
  plasma aldosterone concentration at 8：00 am and 10：00 am
Confirmatory test of primary aldosteronism（Captopril test） | 1 day
  plasma renin concentration at 8：00 am and 10：00 am
circadian cortisol rhythm | 1 day
  adrenocorticotropic hormone at 8：00am、16：00pm and 0：00am
circadian cortisol rhythm | 1 day
  Plasma cortisol concentration at 8：00am、16：00pm and 0：00am
Cortisol metabolism | 1 day
  24-hours urine free cortisol
1 mg (overnight) dexamethasone suppression test | 1 day
  Plasma cortisol concentration at 8：00am
Other indicators of adrenal function | 1 day
  24h urinary，plasma catecholamines and their metabolites
24-hour urine electrolytes | 1 day
  24-hour urine potassium
Imaging of adrenal adenoma | 1 day
  unenhanced and contrast-enhanced CT of adrenal

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Endocrinology, Drum Tower Hospital affiliated to Nanjing University Medical School, Nanjing, Jiangsu, China